CLINICAL TRIAL: NCT00988793
Title: Randomized Trial of Laparoscopic Versus Open Distal Pancreatectomy in Patients With Pancreatic Disease
Brief Title: Laparoscopic Versus Open Pancreatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol needed major revisions; lack of money to institute changes
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0908-05
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic distal pancreatectomy (Active Comparator): Comparison between two different types of surgery, open vs. laparoscopic distal pancreatectomy
  Interventions: Procedure: Laparoscopic distal pancreatectomy
- Open distal pancreatectomy (Active Comparator): Comparison between two different types of surgery, open vs. laparoscopic distal pancreatectomy
  Interventions: Procedure: Open distal pancreatectomy

INTERVENTIONS:
Procedure: Laparoscopic distal pancreatectomy — Comparison of two different types of surgery, laparoscopic versus distal pancreatectomy
  Arms: Laparoscopic distal pancreatectomy
Procedure: Open distal pancreatectomy — Comparison of two different types of surgery, open versus laparoscopic distal pancreatectomy.
  Arms: Open distal pancreatectomy

SUMMARY:
The study will randomized patients to either open or laparoscopic pancreatic surgery. The primary purpose of the study is to determine whether laparoscopic distal pancreatectomy is associated with improved outcomes compared to open distal pancreatectomy.

DETAILED DESCRIPTION:
Open distal pancreatectomy with or without splenectomy has been commonly employed for the treatment of a variety of pancreatic diseases. Although many general surgical procedures have been increasingly performed laparoscopically or with laparoscopic assistance, until the current decade, laparoscopic pancreatic surgery had not been performed. Surgeons at Indiana University Hospital have safely applied laparoscopic surgery to very select patients with pancreatic disease since 2003. Recently, the outcomes of laparoscopic distal pancreatectomy at Indiana University in combination with multiple other institutions were reviewed and presented at the American Surgical Association Meeting 2008. These data suggest that laparoscopic when compared with open distal pancreatectomy may be associated with lower blood loss (357 vs. 588 cc, p<0.01), fewer complications (40 vs. 57%, p<0.01), and shorter hospital stays (5.9 vs. 9.0 days, p<0.01). Furthermore, the laparoscopic approach was an independent predictor of shorter hospital stays. The main criticism of this retrospective study and similarly designed studies is that there is likely to be a selection bias in patients who undergo laparoscopic distal pancreatectomy which may account for the apparent positive results in favor of laparoscopic distal pancreatectomy. In other words, patient factors, not the operative approach may be more predictive of the outcome.

Based on these data, however, laparoscopic distal pancreatectomy appears to be at least as safe as open distal pancreatectomy. Currently, either technique is considered the "standard of care" at Indiana University Hospital as well as several other institutions in the US with expertise in laparoscopic pancreas surgery. To determine whether laparoscopic distal pancreatectomy is truly superior to open distal pancreatectomy in terms of outcomes, we have proposed to randomize patients to laparoscopic vs open distal pancreatectomy. In addition to the randomization, patients will be preoperatively stratified according to whether there is a diagnosis of pancreatic adenocarcinoma, so outcomes in this specific group of patients may be examined. Patients with adenocarcinoma will be randomized separately to insure equal groups in laparoscopic and open distal pancreatectomy groups for this specific diagnosis. Patients with neuroendocrine/islet cell tumors will also be randomized separately to insure equal groups in laparoscopic and open distal pancreatectomy groups for this specific diagnosis. Laparoscopic distal pancreatectomy for adenocarcinoma and neuroendocrine/islet cell tumors is uncommon (e.g., only 9 adenocarcinomas in last 5 years were performed laparoscopically at IU), thus it is clear from the outset that conclusions will be limited about patients with these diagnoses. Although this is being submitted as a single institution study, it will be strongly considered for multi-institutional study design in the near future. Patients will be enrolled on an intention-to-treat manner. Thus, patients who are randomized to laparoscopic distal pancreatectomy who require conversion to open pancreatectomy will still be included in the laparoscopic group in the overall comparative analyses. Subgroup analyses, however, will also be performed excluding this cross-over group.

Objectives:

Primary: The primary objective is to determine whether laparoscopic distal pancreatectomy is associated with improved outcomes compared to open distal pancreatectomy. Retrospective data suggests that blood loss, overall complication rate and hospital length of stay are positively influenced by the laparoscopic approach. Thus, these specific outcomes will be examined:

1. estimated blood loss
2. overall complication rate
3. hospital length of stay

Secondary:

1. to determine whether laparoscopic distal pancreatectomy is safe in patients with pancreatic adenocarcinoma
2. to establish a distal pancreatectomy registry

ELIGIBILITY:
Inclusion Criteria:

* All patients who are eligible for open distal pancreatectomy are also eligible for laparoscopic distal pancreatectomy. There are no absolute contraindications. The only situations where a patient is ineligible is if he/she prefers one approach over the other or the individual surgeon prefers one approach over the other.

NOTE: Patients in whom there is a suspicion of a high likelihood of metastatic pancreatic cancer (minority of patients on trial) will undergo a diagnostic laparoscopy. If the tumor is metastatic (not confined to the pancreas) then the patient is no longer a candidate for any distal pancreatectomy (or the trial). The procedure of diagnostic laparoscopy in this setting is a potential confounder of a trial that randomizes patients to laparoscopic versus open distal pancreatectomy. Due to the importance of cancer patients to this trial, instead of excluding patients from randomization simply because they are undergoing laparoscopy, we have set some limits on the diagnostic laparoscopy. The limits include the use of 2 laparoscopic ports (total) and the diagnostic laparoscopy must be performed at the same setting as the distal pancreatectomy. Thus, after randomization to open distal pancreatectomy, if a patient goes to the operating room, the patient may undergo diagnostic laparoscopy with these limits (2 ports, same setting surgery) prior to undergoing open distal pancreatectomy. This is not an issue with a patient who is randomized for laparoscopic distal pancreatectomy, since when the patient goes to the operating room for diagnostic laparoscopy, they may be transitioned into laparoscopic distal pancreatectomy which allows 5 ports total.

* Patients will be eligible for enrollment in the study if they have a pancreas disease or condition for which they are to undergo distal pancreatectomy. Indications for distal pancreatectomy will be determined by the surgeon caring for the patient.
* Patients must undergo informed consent for the study prior to surgery.
* Patients must be eligible to undergo both open or laparoscopic distal pancreatectomy at all times up until randomization occurs.
* Female patients of child-bearing age must have a negative urine or serum pregnancy test prior to enrollment.
* Patients randomized to laparoscopic technique who require conversion to open technique will remain on trial due to the intention-to-treat design of the study.

Exclusion Criteria:

* Patients who despite pancreas disease or condition are not fit surgical candidates and thus will not undergo distal pancreatectomy.
* Patients who fail to be eligible to undergo both open or laparoscopic distal pancreatectomy at anytime up until randomization occurs.
* Patients undergoing total pancreatectomy.
* Patients undergoing distal pancreatectomy who have had previous right-sided pancreatic resection (i.e., pancreaticoduodenectomy)
* Failure to sign informed consent.
* Pediatric patients (<18 years of age) are excluded from this study.
* Patients who are pregnant.
* Patients with extensive pancreatitis or peri-pancreatic inflammation have a relative contraindication.
* Patients with portal or sinistral hypertension have a relative contraindication.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine whether laparoscopic distal pancreatectomy is associated with improved outcomes compared to open distal pancreatectomy. | 8 months to 5 years

SECONDARY OUTCOMES:
To determine whether laparoscopic distal pancreatectomy is safe in patients with pancreatic adenocarcinoma | 8 months to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Schmidt, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States